CLINICAL TRIAL: NCT02544581
Title: Preliminary Analysis of the Soberlink Alcohol Breath Analyzer System's (SABA) Clinical Utility During Aftercare
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: SoberLink, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mandated impaired professionals: Physicians and other licensed healthcare professionals in mandated monitoring programs by State licensing boards due to Alcohol Use Disorder who are treated with Soberlink combined with aftercare services following residential treatment.
  Interventions: Other: Soberlink combined with aftercare services
- Non-mandated adults: A general population of adults in aftercare following residential treatment for Alcohol Use Disorder who are treated with Soberlink combined with aftercare services following residential treatment.
  Interventions: Other: Soberlink combined with aftercare services

INTERVENTIONS:
Other: Soberlink combined with aftercare services — Soberlink Alcohol Breath Analyzer System combined with aftercare services

SUMMARY:
This is an exempt, retrospective study of a limited set of information obtained from patients' medical records at 10 to 12 substance abuse treatment programs combined with alcohol breath analyzer results during up to 3 years of aftercare monitoring. The study objectives are 1) to compare the compliance rates and likelihood of achieving sustained sobriety for aftercare patients in mandated (eg, impaired professionals) versus non-mandated monitoring programs and 2) identify components within patients' monitoring agreements that are significantly correlated with positive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults with a diagnosis of alcohol abuse enrolled into an aftercare program following residential treatment

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alcohol abusers enrolled into an aftercare program following residential treatment for alcohol abuse
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Compliance rates (negative versus positive versus false positive alcohol test findings) | Test administered 2 to 4 times per day for up to 3 years
Response rates: defined as use of device when prompted-will include several values such as missed, late, excused | Test administered 2 to 4 times per day for up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ed Pigott, Ph.D., Principal Investigator — Mr. Pigott
Locations (1):
- Ed Pigott, Juno Beach, Florida, United States